CLINICAL TRIAL: NCT05826678
Title: A Pilot Clinical Trial to Assess Feasibility, Facilitators and Barriers of Continuous Glucose Monitoring in Asian Americans With Type 2 Diabetes
Brief Title: Trial to Assess Continuous Glucose Monitoring in Asian Americans With Type 2 Diabetes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Joslin Diabetes Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: STUDY00000206
Record Dates: First submitted 2023-04-12; First posted 2023-04-24 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Continuous Glucose Monitoring; Health Disparity
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Participants on CGM (Active Comparator): Participants in this group will be offered a CGM device for glucose monitoring, with training and educational materials provided in either English or Chinese, according to the participant's preference.
  Interventions: Device: Continuous Glucose Monitor
- Participants on Finger-stick only (Placebo Comparator): Participants in this group continue standard fingerstick self-monitoring of blood glucose (FSGM) as per standard care protocol. They will also receive educational materials provided in either English or Chinese, according to the participant's preference.
  Interventions: Behavioral: Finger stick glucose monitoring

INTERVENTIONS:
Device: Continuous Glucose Monitor — The Clinical Diabetes Educator (CDE) will follow up with the participants at Month 1 after the baseline study visit, at the study midpoint (Month 3), and at the end of the study (Month 6) to check CGM usage, including timely calibration and change adherence. At the end of the study, participants will be invited to complete a survey and participate in virtual interviews to assess changes in their health behaviors and the acceptability of CGM devices.
  Arms: Participants on CGM
Behavioral: Finger stick glucose monitoring — Participants will adhere to the standard care protocol and continue self-monitoring of blood glucose through fingersticks as per usual practice[46]. The Clinical Diabetes Educator (CDE) will monitor and provide follow-up to the control group participants as per the same schedule followed for the intervention group.
  Arms: Participants on Finger-stick only

SUMMARY:
This study aims to understand the use of continuous glucose monitors (CGM) in Asian Americans with type 2 diabetes (T2D). Researchers will compare participants on continuous glucose monitors with participants using fingerstick self-monitoring with the aim of answering the following questions:

1. Check if continuous glucose monitoring is doable and consistent for this group, and see how it affects their quality of life.
2. Estimate how well the health outcomes (glucose and lipid markers) vary over the study period.
3. Understand how social and community factors can impact the use of continuous glucose monitors in this group.

DETAILED DESCRIPTION:
The Type 2 Diabetes (T2D) pandemic continues to expand in the U.S. and globally. However, the prevalence of T2D is much higher in Asian-Americans (AA) and in other minorities compared to non-Hispanic Whites in the U.S, and AAs have the highest age- and sex-adjusted undiagnosed rate of T2D (7.5%) compared to all other ethnic and racial groups. There is ample evidence that disparities in diagnosis and care for T2D exist in AA communities. The majority of AAs are 1st generation immigrants, and this has further contributed to the disparity in care and diagnosis of diabetes due to the following reasons:

1. Higher unawareness rate: A major contributor to higher T2D unawareness among AAs is the significant difference in BMI-associated T2D risk among AAs (24-25 kg/m2) compared with non-Asians (29-30 kg/m2). Until the "Screen at 23" campaign (See "Innovation"), no national agency would recognize and recommend that AAs be screened for T2D at lower BMIs of 23-25 kg/m2. Furthermore, NHANES data has shown that while age- and sex-adjusted diabetes prevalence among AAs is 19%, the breakdown of this figure may not be truly reflective of the actual prevalence among the disaggregated AA subgroups, which showed a wide variation with South Asians at 23%, Southeast Asians at 22%, and East Asians (including Chinese, Koreans and Japanese) at 14%, the last one being comparable to a recent report from China which showed diabetes prevalence of 11.2%.
2. Cultural and language barriers: AAs living in the US have the highest rates (35%) of limited English proficiency. This figure is even higher at 44% for foreign-born ChA. Limited English proficiency is closely linked to reduced health access, poor health outcomes and lower utilization rates of health technologies.
3. Model minority myth: Hurdles to health care have been significantly exacerbated by the exponential rise in anti-Asian sentiments during the COVID-19 pandemic.

Rapidly advancing diabetes technologies, especially CGM, can achieve better metabolic targets, lower diabetes-related complications, and provide a better quality of life, which have been reported for other ethnic groups but not for AAs due to the systemic exclusion of AAs from CGM studies. Multiple systemic barriers exist for AA to access CGMs, including costs and lack of data to justify reimbursement, provider inertia, and lack of advocacy and vocalization of needs, on top of limited English proficiency and lack of culturally-tailored education. These barriers are in addition to a lack of "Digital Literacy", the new "super social determinant of health", which will increase disparities between those who have skills and access to digital tools and those who do not. In this proposal, we will evaluate the impact, barriers and facilitators of CGM use and adherence in AAs (1st generation ChA) with T2D.

In this 6-month clinical trial, we will examine the impact of CGM use vs. No CGM among 1st generation ChA with T2D.The aim will be to:

1. Evaluate feasibility (adherence and consistency) and quality of life measures during CGM use in this population.
2. Generate precision estimates of the distribution of the secondary outcomes (6-month glycemic control and lipid markers) in both arms to inform a future randomized controlled trial (RCT).

3: Identify multi-level barriers and facilitators of CGM use for ChA with T2D, using a socioecological framework (patient-level, provider-level, and community/environment level). We aim to comprehensively evaluate the implementation process (facilitators and impediments), resource requirements, and intermediate patient adherence outcomes for the program using mixed-methods approaches. These will inform the design of culturally-tailored interventions for larger RCT.

ELIGIBILITY:
Inclusion Criteria:

* Chinese Americans 40 years and older who are 1st generation immigrants, currently residing in the US, and clinically diagnosed with T2D.
* CGM-naïve
* HbA1c >7.5% within 3 months of study commencement.
* Participants should also possess a smartphone, as this is needed in order to facilitate the collection of CGM data by the study team as well as homogenize CGM usage education.

Exclusion Criteria:

* Known diagnosis of dysfunction/dementia or learning disabilities
* Not fluent in either English or Chinese
* Currently undergoing or planning to undergo diathermy or high-frequency heat treatments in whom CGM use may be contraindicated
* Inability to travel due to frailty or health reasons
* Lack of internet access
* Critically ill populations, including those on dialysis
* Vulnerable populations (prisoners and women who are pregnant or planning to be pregnant during the time of study)

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-09-22 (Actual); Primary Completion 2024-05-15 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility (CGM device adherence) | 6 month
  Number of hours device is active in total for the entire 6 month study period
Feasibility (Consistency) 1 | 6 months
  Proportion CGM program elements completed at each visit against a checklist of pre-specified essential elements
Feasibility (Consistency) 2 | 6 months
  Average session duration as compared to assigned time plan.
World Health Organization (Five) Well-Being Index (WHO-5) change over 6 month study period | Change in measure comparing Baseline and 6 months
  WHO-5 uses a five-item scale to assess overall well-being
EQ-5D-5L change over 6 month study period | Change in measure comparing Baseline and 6 months
  EQ-5D-5L assesses health status both as an overall self-rated health on a visual analog scale and across five areas (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) with three levels of severity (no/mild, moderate, or severe problems)
Diabetes Distress Scale (DDS) change over 6 month study period | Change in measure comparing Baseline and 6 months
  DDS is a 17-item scale that measures worry and concerns specifically related to diabetes and its management
Hypoglycemic Confidence Scale (HCS) change over 6 month study period | Change in measure comparing Baseline and 6 months
  HCS is a nine-item survey that evaluates the degree to which patients feel able, secure, and comfortable about their ability to stay safe from hypoglycemic-related problems

SECONDARY OUTCOMES:
HbA1c change (%) from 0-6 months | Change in measure comparing Baseline and 6 months
  HbA1c change (%) between baseline (0 months) and end of intervention period (6 months) will be assessed as a continuous response variable for each study arm
Time in range (TIR) metrics change (%) from 0-6 months | Change in measure comparing Baseline and 6 months
  Change in %TIR metrics between baseline (0 months) and end of intervention period (6 months) will be assessed as a continuous response variable for the CGM+ arm
Lipid changes from 0-6 months | Change in measure comparing Baseline and 6 months
  We plan to assess the changes from baseline to 6 months for levels of lipid profile components, including total cholesterol, triglyceride, low-density lipoprotein (LDL), and high-density lipoprotein (HDL) levels.
Blood pressure changes from 0-6 months | Change in measure comparing Baseline and 6 months
  We will assess change from baseline to 6 months for systolic and diastolic blood pressures.
eGFR changes from 0-6 months | Change in measure comparing Baseline and 6 months
  We will assess change from baseline to 6 months for eGFR
Diabetes Knowledge and Behavior change from 0-6 months | Change comparing Baseline and 6 months
  Assessed through Semi-structured virtual interviews that will be conducted at the Baseline and 6-month mark.
Family/social-level factors impacting technological device for care management | Change comparing Baseline and 6 months
  Semi-structured virtual interviews conducted at baseline and 6-month mark (in both arms) will also probe participants on broad topics of stigmas related to technology will be assessed with more directed questions on stigmas in varying environments-home, work, and in social gatherings.

CONTACTS AND LOCATIONS:
Overall Officials: George King, MD, Principal Investigator — Joslin Diabetes Center
Locations (1):
- Joslin Diabetes Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided